CLINICAL TRIAL: NCT02189798
Title: Implantation of the HiRes90K™ Advantage Cochlear Implant With HiFocus™ Mid-Scala and Development of a Combined Electric and Acoustic Stimulation Technology in Adults With Partial Deafness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Thirty-five subjects wore the EAS processor for as long as 84 months without significant safety issues. Sufficient data gained to support EAS technology development for safe use in subjects with residual low-frequency acoustic hearing sensitivity.
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR0114
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss; Partial Deafness; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases
Keywords: Cochlear Implant; HiRes™ 90K Advantage implant; Cochlear Implantation; HiFocus™ Mid-Scala electrode; Listening Benefits; Adults; Cochlear Implant Benefit; Electrical Stimulation; Electro-Acoustic Stimulation (EAS)
MeSH Terms: conditions — Hearing Loss; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases

STUDY DESIGN:
Intervention Model Description: The two main arms are conducted in parallel. The third arm is optional for subjects who complete either of the two main arms using the EAS sound processor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Newly Implanted Group (Experimental): HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with partial deafness. Patients retaining considerable low frequency acoustic hearing after the surgery, will be fitted with the EAS sound processor.
  Interventions: Device: HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode; Device: EAS sound processor
- Existing Implanted Group (Experimental): Adults unilaterally implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode with partial deafness will be fitted with the EAS sound processor.
  Interventions: Device: EAS sound processor
- EAS Extended Use Arm (Experimental): Adults who are unilaterally implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode with partial deafness and completed the 12 Month visit using the EAS sound processor in either the Newly Implanted Group or Existing Implanted Group.
  Interventions: Device: EAS sound processor

INTERVENTIONS:
Device: HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode — HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss).
  Arms: Newly Implanted Group
Device: EAS sound processor — Patients with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss) implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be fitted with the EAS sound processor.

SUMMARY:
The purpose of this feasibility study is to evaluate whether low-frequency acoustic hearing sensitivity can be preserved in newly implanted adults with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss) using the HiResolution™ 90K™ Advantage cochlear implant with the HiFocus™ Mid-Scala electrode to support the development of electro-acoustic stimulation technology (EAS).

ELIGIBILITY:
Inclusion criteria: Newly Implanted Group:

* Ability to provide informed consent
* No previous cochlear implant experience in either ear
* 18 years of age or older
* Up to a moderate sensorineural hearing loss in the low-to-mid frequencies (pure tone average ≤65 dB for 125, 250, 500, and 1000 Hz) and a severe-to-profound sensorineural hearing loss in the high frequencies (pure tone average ≥ 70 dB HL for 2,000, 3000, 4,000, and 8,000 Hz) in the ear to be implanted
* Aided CNC word recognition score up to 50% in ear to be implanted
* Up to a moderate sensorineural hearing loss in the low-to-mid frequencies (pure tone average ≤65 dB for 125, 250, 500, and 1000 Hz) and a severe-to-profound sensorineural hearing loss in the high frequencies (pure tone average ≥ 70 dB HL for 2,000, 3000, 4,000, and 8,000 Hz) in the contralateral (non-implanted) ear
* Aided CNC word recognition score up to 80% in the contralateral ear
* English language proficiency
* Willingness to use an ear-level sound processor postoperatively for the duration of the study trial
* Willingness to participate in all scheduled procedures outlined in the protocol

Exclusion Criteria: Newly Implanted Group:

* Preoperative audiometric conductive overlay of 15 dB or greater at two frequencies or more in range of 500-1000 Hz in the ear to be implanted
* Congenital hearing loss (for purpose of this study, onset prior to age 2 years*). *Based on critical period for speech and language development
* Duration greater than 30 years of severe-to-profound high-frequency hearing loss
* Cochlear malformation or obstruction that would preclude full insertion of electrode array in the ear to be implanted
* Medical or psychological conditions that contraindicate surgery or impact the ability to manage an implanted device or the study related procedures as determined by the investigator
* Deafness due to central auditory lesion or cochlear nerve deficiency, diagnosis of auditory neuropathy/dys-synchrony in either the ear to be implanted or the contralateral ear
* Active middle-ear disease/infection in the ear to be implanted
* Unrealistic expectations regarding potential benefits, risks and limitations inherent to implant surgical procedures as determined by the investigator
* Unwillingness or inability of subject to comply with all investigational requirements as determined by the investigator

EAS Fitting Inclusion Criteria: Newly Implanted and Existing Implanted Groups

* Ability to provide informed consent
* 18 years of age or older, unilaterally implanted with HiRes90K™ Advantage cochlear implant with HiFocus™ Mid-Scala electrode and fit with an ear-level sound processor (i.e. Naída family device)
* Postoperative unaided low frequency audiometric hearing thresholds in the treated ear up to 80 dB HL for at least one frequency from 125 - 1000 Hz
* English Language Proficiency
* Willingness to participate in all scheduled procedures outlined in the study protocol

EAS Fitting Exclusion Criteria: Newly Implanted and Existing Implanted Groups

* Unilaterally implanted with HiRes 90K™ Advantage cochlear implant with HiFocus™ Helix® and HiFocus™ 1j electrode
* Exclusive use of a body worn external sound processor
* Deafness due to central auditory lesion or cochlear nerve deficiency, diagnosis of auditory neuropathy/dys-synchrony in either the implanted or the contralateral ear
* Postoperative unaided low frequency audiometric hearing thresholds in the treated ear exceeding 80 dB HL at each frequency from 125 - 1000 Hz Unwillingness or inability of subject to comply with all investigational requirements as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Tampa Bay Hearing and Balance Center, Tampa, Florida
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Midwest Ear Institute/St. Luke's Health System, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Oklahoma Ear Institute, Oklahoma City, Oklahoma
  - Vanderbilt Bill Wilkerson Center, Nashville, Tennessee
  - Austin Ear, Nose & Throat Clinic, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators recruited study subjects from their clinical practices. Thirteen study sites enrolled a total of 67 subjects. Of those enrolled, 35 completed the study main phase (month 12). The first patient first visit occurred on June 30, 2014, and last patient last visit occurred on 11/2/2020 for the main phase of the study. Twenty-four of the subjects that completed month 12 volunteered to enroll in the extended use phase. The last visit of the extended use phase was March 29, 2022.
Period: Main Phase
Arm/Group | Newly Implanted Group | Existing Implanted Group
Started | 49 | 18
Completed | 22 | 13
Not Completed | 27 | 5
Period: Extended Use Phase
Arm/Group | Newly Implanted Group | Existing Implanted Group
Started | 15 (Participation in the Extended Use phase is voluntary after completion of Main Phase month12 visit.) | 9 (Participation in the Extended Use Phase if voluntary after completion of the Main Phase month 12 visit.)
Completed | 0 | 0
Not Completed | 15 | 9
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Desire to explore other commercial technology/Processor Upgrade | 11 | 1
Not completed — Explanted prior to 24 month visit | 1 | 0
Not completed — Travel Issues | 2 | 1
Not completed — No longer perceiving a benefit from acoustic component | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly Implanted Group | Existing Implanted Group | Total
Number analyzed (Participants) | 49 | 18 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 12 | 35
  >=65 years | 26 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13.95) | 60.3 (12.37) | 64 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 6 | 33
  Male | 22 | 12 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 18 | 67
Unaided low frequency hearing threshold - EAS Baseline [Mean (Standard Deviation); unit: Hertz (Hz)] — Population: Low-frequency pure tone hearing ability (250-1000 Hz) was tested by playing tones and measuring the softest sounds the subject could hear. For EAS eligibility, candidates needed to hear at least one low-frequency tone at 80 dB HL or better after surgery without a hearing aid. Only those who met this criterion, used the investigational device, and completed the main EAS phase were included in the analysis.
  Hertz (Hz)
    number analyzed (Participants) | 15 | 10 | 25
    (all) | 67 (11) | 72.0 (19.5) | 69 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Unaided Pure-tone Average (PTA) Hearing Threshold Measurements
Description: Unaided pure tone hearing threshold measurement in the implanted ear at months 3, 6 and 12 months after surgery compared to pre-implant audiometric thresholds (using pure-tone average of 125 - 1000 Hz for comparison)
Time Frame: Twelve months post device activation
Population: Analysis includes only subjects who completed up to month 3 using the EAS processor.
Measure: Mean (Standard Deviation); unit: decibles
Groups:
- Newly Implanted Subjects: HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with partial deafness. Patients retaining considerable low frequency acoustic hearing after the surgery, were fitted with the EAS sound processor.
  HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode: HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss).
  EAS sound processor: Patients with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss) implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be fitted with the EAS sound processor.
- Existing Implanted: Adults unilaterally implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode with partial deafness will be fitted with the EAS sound processor.
  EAS sound processor: Patients with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss) implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be fitted with the EAS sound processor.
Arm/Group | Newly Implanted Subjects | Existing Implanted
Number analyzed (Participants) | 15 | 10
decibles
  Baseline PTA | 46.7 (8.7) | 72.0 (19.5)
  3 Month PTA | 69.4 (12.1) | 71.6 (20.5)
  6 Month PTA | 67.5 (12.2) | 72.6 (18.9)
  12 Month PTA | 71.6 (15.6) | 74.5 (17.1)

2. Primary Outcome: Consonant-Nucleus-Consonant (CNC) Word Recognition Test in Quiet
Description: Consonant-Nucleus-Consonant (CNC) Word Recognition Test in quiet in the treated ear measured at Month 1, 3, 6 and 12 post device activation compared to pre-implant speech perception testing in quiet. Scores are determined on scale of 0% to 100% words correct with higher scores indicating a better outcome.
Time Frame: Up to 12 months post device activation
Population: Analysis includes only subjects who completed up to month 12 using the EAS processor.
Measure: Mean (Standard Deviation); unit: Percent words correct
Groups:
- Newly Enrolled: HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with partial deafness. Patients retaining considerable low frequency acoustic hearing after the surgery, will be fitted with the EAS sound processor.
  HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode: HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss).
  EAS sound processor: Patients with partial deafness (considerable low frequency acoustic hearing profiles with severe-to-profound high frequency sensorineural hearing loss) implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be fitted with the EAS sound processor.
Arm/Group | Newly Enrolled | Existing Implanted
Number analyzed (Participants) | 15 | 10
Percent words correct
  Baseline | 19.3 (13.5) | 61.5 (19.5)
  Month 1 Post Device /EAS Activation | 31.3 (25.8) | 67.1 (17.8)
  Month 3 Post Device /EAS Activation | 50.4 (28.0) | 70.5 (15.9)
  Month 6 Post Device /EAS Activation | 50.5 (25.6) | 72.7 (18.3)
  Month 12 Post Device /EAS Activation | 51.1 (25.0) | 73.3 (19.2)

3. Primary Outcome: Speech Perception Testing (AzBio) in Noise.
Description: Speech perception testing (AzBio) in noise in the treated ear measured at Month 1, 3, 6 and 12 post device activation compared to pre-implant speech perception testing in quiet. Scores are determined on scale of 0% to 100% words correct with higher scores indicating a better outcome.
Time Frame: up to 12 months post device activation
Population: Analysis includes only subjects who completed the main phase study using the EAS processor.
Measure: Mean (Standard Deviation); unit: Percent words correct
Arm/Group | Newly Enrolled | Existing Implanted
Number analyzed (Participants) | 15 | 15
Percent words correct
  Baseline | 11.9 (8.5) | 46.2 (22.6)
  1 Month Post Device/ EAS Activation | 19 (19.7) | 55.0 (27.1)
  3 Month Post Device/ EAS Activation | 42.1 (28.3) | 57.7 (25.8)
  6 Month Post Device/ EAS Activation | 44.4 (28) | 62.6 (27.1)
  12 Month Post Device/ EAS Activation | 46.2 (26.3) | 64.1 (23.2)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were documented from the signing of the informed consent form through two weeks after the final study visit, up to 12 months post-activation in the main phase. In the extended use phase, participants were assessed annually, with AEs tracked as reported until exit. The first subject exited at 24 months, while the last exited at 84 months post-device activation.
Description: Information recorded includes onset date, if the AE is serious, categorization, description, course of action taken, status, and relation to study device or procedure. The number subjects experiencing AEs will be summarized by type and frequency of event.
Groups:
- Extended Use Phase - Newly Implanted Group: Adults who are unilaterally implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode with partial deafness and completed the 12 Month visit using the EAS sound processor in the Newly Implanted Group.
  Enrollment was optional and subject to the willingness of the participant and the discretion of the managing clinician.
- Extended Use Phase - Existing Implanted Group: Adults who are unilaterally implanted with HiRes 90K™ Advantage implant with HiFocus™ Mid-Scala electrode with partial deafness and completed the 12 Month visit using the EAS sound processor in the Existing Implanted Group.
  Enrollment was optional and subject to the willingness of the participant and the discretion of the managing clinician
Arm/Group | Newly Implanted Group | Existing Implanted Group | Extended Use Phase - Newly Implanted Group | Extended Use Phase - Existing Implanted Group
All-Cause Mortality (participants affected / at risk) | 1/49 | 0/18 | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 16/49 | 0/18 | 1/15 | 0/9
Other Adverse Events (participants affected / at risk) | 24/49 | 9/18 | 4/15 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Newly Implanted Group (N=49) | Existing Implanted Group (N=18) | Extended Use Phase - Newly Implanted Group (N=15) | Extended Use Phase - Existing Implanted Group (N=9)
Severe inflammation from extensive radiation damage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject hospitalized for treatment.
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject passed away in their sleep. Event reported by subject's spouse.
Fractured left femoral head secondary to fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject hospitalized for treatment.
Fractured rib secondary to fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject hospitalized for treatment.
Crushed legs secondary to Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject hospitalized for treatment.
Hospitalization due to Health Setback (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject hospitalized
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Subject hospitalized
Complication at Implant Site (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Torn Shoulder Tendon (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Required Surgical Repair
Postoperative decrease/loss of residual hearing (Ear and labyrinth disorders) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Newly Implanted Group (N=49) | Existing Implanted Group (N=18) | Extended Use Phase - Newly Implanted Group (N=15) | Extended Use Phase - Existing Implanted Group (N=9)
Condition of the Contralateral ear (Ear and labyrinth disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Complication at Implant site (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Oral/Taste disturbance (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased Concentration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related/ Programming Problems (Product Issues) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Irritation/Pain (Ear and labyrinth disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
External/Middle Ear Postoperative Symptom (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye Fluttering - Right eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headaches (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Iron Deficiency/Low Hemoglobin count
Leaky Heart Valve (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lockjaw with pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular Degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal injury, sprain or fracture (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 0 (0) | 0 (0)
Numbness (Implanted Ear) (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral/Dental Disturbance (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pain due to bone fracture from a fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative decrease/loss of residual hearing (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea after implant surgery in contralateral ear (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-operative Pain - Implanted ear (Surgical and medical procedures) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Postoperative popping noise (Implanted Ear) (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative Sensation of clogged ear (Implanted Ear) (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Postoperative Sensitivity during testing (Implanted Ear) (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prediabetes (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostate Dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal illness (injury, stones or failure) (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin irritation - Implant site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (General) (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 1 (1) | 0 (0)
Sleep Deprivation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somatosensory response to sound at certain frequencies (Bilateral) (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Uterine Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical Complication - Implanted Ear (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste Disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus - Implanted Ear (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Tinnitus - Contralateral Ear (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinnitus - Continuous (Bilateral) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo or Dizziness (Ear and labyrinth disorders) | 12 (16) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02189798/Prot_SAP_000.pdf